CLINICAL TRIAL: NCT06524999
Title: The Effect of Progressive Muscle Relaxation Exercises on Vital Signs, Anxiety And Comfort Level of Patients Undergoing Coronary Angiography
Brief Title: Effect of Progressive Muscle Relaxation on Anxiety and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Tuğçe Türten Kaymaz, Assist. Prof., Ankara Yildirim Beyazıt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AnkaraYBU-SBF-TTK-02
Record Dates: First submitted 2024-07-19; First posted 2024-07-29 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-08

CONDITIONS: Muscle Relaxation; Coronary Artery Disease
Keywords: Anxiety; coronary angiography; patient comfort; progressive relaxation exercise; vital signs
MeSH Terms: conditions — Coronary Artery Disease; Anxiety Disorders | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Progressive muscle relaxation (Experimental): The researcher provided the intervention group participants face-to-face training on progressive relaxation exercises (PREs) at the first hospitalization. She had developed "A Guide to Progressive Relaxation Exercises" based on a literature review. The guide consisted of 22 steps. After the briefing, the researcher asked each intervention group participant to perform the PREs with voice instructions. The study continued with participants who performed the PRE steps correctly. While the participant was performing PREs, the researcher guided her verbally in line with the guide. After the nurse teaches the PRE technique once, the individual can apply it.
  Progressive relaxation exercises are performed for about 15-30 minutes.
  Interventions: Behavioral: Progressive muscle relaxation
- Control (No Intervention): In this group, participant were assessed without any other intervention.

INTERVENTIONS:
Behavioral: Progressive muscle relaxation — This intervention consists of two parts. The first part gives short information about the content and how exercises should be done. It consists of information about deep relaxation. In the second part, there are relaxation exercises accompanied. Both the briefing and the intervention lasted 30 minutes for each patient.
  Arms: Progressive muscle relaxation

SUMMARY:
This study aimed to examine the effect of relaxation exercise applied to patients who will undergo elective coronary angiography (CAG) for the first time, on their vital signs, anxiety and comfort levels.

The main questions it aims to answer are:

1. Does progressive relaxation exercises affect CAG patients' vital signs.
2. Does progressive relaxation exercises affect CAG patients' anxiety levels.
3. Does progressive relaxation exercises affect CAG patients' comfort levels. Researchers will compare the intervention group with the control group to see if relaxation exercise is effective.

Before coronary angiography, patients will undergo a relaxation exercise once. Vital signs, comfort and anxiety level will be evaluated before and after angiography.

DETAILED DESCRIPTION:
Coronary angiography (CAG) is considered the "gold standard" in determining coronary anatomy. And it is used very frequently in the diagnosis and treatment of coronary artery disease. CAG, which is an invasive procedure, causes anxiety in patients undergoing the procedure. Anxiety leads to negative consequences in vital signs such as increased blood pressure, pulse and respiration rate, and pain intensity. Pain, anxiety and many factors that develop due to invasive procedures such as angiography also reduce the comfort level of patients. Reducing anxiety and pain, preventing negativities in vital signs, and increasing comfort contribute to the success of the procedure, the patient's level of well-being, and satisfaction with health care services. This study aimed to determine the effect of progressive relaxation exercise on patients' vital signs, anxiety and comfort levels in patients undergoing angiography.

ELIGIBILITY:
Inclusion Criteria:

* undergo CAG for the first time
* has a chest score of 5 or less on the pain scale
* has no history of mental disorder according to medical records
* is able to communicate

Exclusion Criteria:

* Admission to the intensive care unit after the CAG procedure
* starting analgesic or perlinganit infusion
* wanting to quit the research

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
State Anxiety Scale | First assessment; before intervention. Second assessment; immediately after the muscle exercise, immediately before the angiography. Third assessment; approximately 30 minute after the angiography.
  The State Anxiety Scale (SAS) shows how an individual feels under certain circumstances at certain times. It consists of 20 items rated on a four-point Likert-type scale ("1: none" to "4: all"). The total score ranges from 20 to 80, with higher scores indicating more anxiety.

SECONDARY OUTCOMES:
The General Comfort Scale Short Form | First assessment; before intervention. Second assessment; immediately after the muscle exercise, immediately before the angiography. Third assessment; approximately 30 minute after the angiography.
  The General Comfort Scale Short Form assesses how comfortable an individual feels at the moment. The form consists of 28 items rated on a six-point Likert-type scale ("1=strongly disagree" to "6=strongly agree"). The total score ranges from 28 to 168, with higher scores indicating higher levels of comfort.
The Vital Signs Follow-up (for blood pressure) | First assessment; before intervention. Second assessment; immediately after the muscle exercise, immediately before the angiography. Third assessment; approximately 30 minute after the angiography.
  The Vital Signs Follow-up Chart was developed by the researchers to record the parameters of blood pressure.
The Vital Signs Follow-up (for pulse) | First assessment; before intervention. Second assessment; immediately after the muscle exercise, immediately before the angiography. Third assessment; approximately 30 minute after the angiography.
  The Vital Signs Follow-up Chart was developed by the researchers to record the parameters of pulse.
The Vital Signs Follow-up (for respiration) | First assessment; before intervention. Second assessment; immediately after the muscle exercise, immediately before the angiography. Third assessment; approximately 30 minute after the angiography.
  The Vital Signs Follow-up Chart was developed by the researchers to record the parameters of respiration.
The Vital Signs Follow-up (saturation) | First assessment; before intervention. Second assessment; immediately after the muscle exercise, immediately before the angiography. Third assessment; approximately 30 minute after the angiography.
  The Vital Signs Follow-up Chart was developed by the researchers to record the parameters of saturation.
The Vital Signs Follow-up (for body temperature) | First assessment; before intervention. Second assessment; immediately after the muscle exercise, immediately before the angiography. Third assessment; approximately 30 minute after the angiography.
  The Vital Signs Follow-up Chart was developed by the researchers to record the parameters of body temperature.
The Visual Analog Scale | First assessment; before intervention. Second assessment; immediately after the muscle exercise, immediately before the angiography. Third assessment; approximately 30 minute after the angiography.
  The Visual Analog Scale (VAS) is a 10 cm long horizontal or vertical line with anchor statements "no pain or pain at its least" at the left-most end and "unbearable pain or worst pain imaginable" at the right-most end. The VAS is scored on a scale of 0 to 10 (0 = no pain, 1-3 = mild pain, 4-7 moderate pain, 8-10 = severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Tuğçe Türten Kaymaz, PhD, Principal Investigator — Ankara Yildirim Beyazıt University; Beyza Güney, MSc, Principal Investigator — Duzce University Faculty of Medicine Hospital
Locations (1):
- Ankara Yildirim Beyazıt University, Ankara, Çubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No